CLINICAL TRIAL: NCT03523078
Title: Cosmetic Outcome, Patient-reported Outcomes, and Reconstruction-related Complications in Breast Cancer Women Treated With or Without Post-mastectomy Radiation Therapy: Prospective Cohort Study
Brief Title: Cosmetic Outcome, Patient-reported Outcomes, and Reconstruction-related Complications in Breast Cancer Women Treated With or Without Post-mastectomy Radiation Therapy
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Yonsei University (Other)
Responsible Party: Sponsor
Other Study IDs: 4-2017-1108
Record Dates: First submitted 2018-05-01; First posted 2018-05-14 (Actual); Last update posted 2020-09-29 (Actual); Status verified 2020-09

CONDITIONS: Breast Cancer Female

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Procedure: Breast reconstructive surgery — All sorts of breast reconstructive surgery are allowed in this study in terms of timing, autologous/prosthetic and so forth.

SUMMARY:
This study aim to investigate the breast reconstruction outcome after mastectomy with or without radiation therapy from the patient's point of view.

ELIGIBILITY:
Inclusion Criteria:

* Pathologically confirmed invasive breast carcinoma
* Women who underwent mastectomy and breast reconstruction
* Good performance status (ECOG 0-1)

Exclusion Criteria:

* Recurrent breast cancer
* History of ipsilateral breast irradiation

Min Age: 20 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Women undergoing reconstruction surgery after mastectomy at an academic center
Sampling Method: Non-Probability Sample
Enrollment: 500 (Estimated)
Dates: Start 2018-02-01 (Actual); Primary Completion 2024-02-01 (Estimated); Study Completion 2024-02-01 (Estimated)

PRIMARY OUTCOMES:
Change from baseline of Breast-Q questionnaire score | Before mastectomy & reconstruction surgery (allowed up to 8 weeks ago)
  Patient reported outcome measures include psychosocial functioning, patient treatment satisfaction, physical functioning, body image and pain. (Breast-Q survey)
Change from baseline of Breast-Q questionnaire score | Immediate after the last reconstructive procedures/surgery (allowed plus 8 weeks)
  Patient reported outcome measures include psychosocial functioning, patient treatment satisfaction, physical functioning, body image and pain. (Breast-Q survey)
Change from baseline of Breast-Q questionnaire score | 1 year after the last reconstructive procedures/surgery (allowed plus 8 weeks)
  Patient reported outcome measures include psychosocial functioning, patient treatment satisfaction, physical functioning, body image and pain. (Breast-Q survey)

SECONDARY OUTCOMES:
Reconstruction complications | within 1 year after last reconstruction procedures (plus 8 weeks)
  Patient reported outcome measures include psychosocial functioning, patient treatment satisfaction, physical functioning, body image and pain. (Breast-Q survey)

CONTACTS AND LOCATIONS:
Locations (1):
- Severance Hospital, Seoul, Korea, South Korea

REFERENCES:
- [Derived] Chung SY, Chang JS, Shin KH, Kim JH, Park W, Kim H, Kim K, Lee IJ, Yoon WS, Cha J, Lee KC, Kim JH, Choi JH, Ahn SJ, Ha B, Lee SY, Lee DS, Lee J, Shin SO, Lee SW, Choi J, Kim MY, Kim YJ, Im JH, Suh CO, Kim YB. Impact of radiation dose on complications among women with breast cancer who underwent breast reconstruction and post-mastectomy radiotherapy: A multi-institutional validation study. Breast. 2021 Apr;56:7-13. doi: 10.1016/j.breast.2021.01.003. Epub 2021 Jan 20. PMID 33517043
- [Derived] Chang JS, Song SY, Oh JH, Lew DH, Roh TS, Kim SY, Keum KC, Lee DW, Kim YB. Influence of Radiation Dose to Reconstructed Breast Following Mastectomy on Complication in Breast Cancer Patients Undergoing Two-Stage Prosthetic Breast Reconstruction. Front Oncol. 2019 Apr 9;9:243. doi: 10.3389/fonc.2019.00243. eCollection 2019. PMID 31024845